CLINICAL TRIAL: NCT04410276
Title: VENOUS: A Translational Study of Enterococcal Bacteremia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Cesar A Arias, Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-15-0055
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Enterococcal Bacteremia
Keywords: entercoccal bloodstream infection; vancomycin-resistant enterococci; vancomycin-susceptible enterococci

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples With DNA — Enterococcal isolates from index and subsequent blood cultures will be collected by the research personnel from the clinical microbiology lab. Bacterial isolates will be processed by conventional laboratory methods at each institution. Isolates will be stored at -80º Celsius using local laboratory standards until shipment to central laboratory (UTHealth) for storage and further characterization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with enterococcal bloodstream infections: Adult patients (≥ 18 years of age) with ≥ 1 positive blood cultures with Enterococcus during hospitalization and who have repeat blood culture(s) within 7 days from the first positive culture will be included.

SUMMARY:
The purpose of this study is to assemble a multicenter prospective cohort of patients with enterococcal bloodstream infections (BSIs) to provide data on outcomes of patients with enterococcal BSIs for sample size calculations for future trials, as well as to characterize enterococcal isolates causing BSIs in order to comprehensively dissect the molecular epidemiology of infecting organisms for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient
* ≥1 positive blood culture with Enterococcus spp. (VRE or VSE) during hospitalization
* bacterial isolate(s) is/are available for further characterization
* Repeat blood culture(s) within 7 days from the first positive culture

Exclusion Criteria:

* Cultures obtained from patients not admitted to the hospital
* Isolate(s) not available for further studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
All-cause, in-hospital mortality | 30 days or until hospital discharge
  Death by any cause while patient is in the hospital

SECONDARY OUTCOMES:
Number of participants with microbiological outcome | 7 days after first documented positive blood culture
  Eradication defined as a negative follow-up blood culture > 4 days after index blood culture
Number of participants with recurrence of bacteremia | 14 days after the documented eradication of bacteremia
  Positive blood culture with the same organism within the following 14 days after the documented eradication of bacteremia

CONTACTS AND LOCATIONS:
Overall Officials: Cesar A. Arias, MD, MSc, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (12):
- United States (8):
  - Jackson Health System, University of Miami Miller School of Medicine, Miami, Florida
  - Henry Ford Hospital and Medical Centers, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Hospital Sanatorio, Buenos Aires, Argentina
- Hospital Padre Hurtado, Santiago, Chile
- University of Cologne, Cologne, Germany
- Hospital Universitari de Bellvitge, Barcelona, Spain